CLINICAL TRIAL: NCT03166189
Title: Open Randomized Trial of Clinical Efficiency and Safety of Cell Product of Autologous Bone Marrow-derived Mesenchymal Stem Cells for Reparative Treatment of Destructively Changed Endometrium in Patients With Repeated IVF Failures
Brief Title: Autologous Bone Marrow-derived Mesenchymal Stem Cells for Atrophic Endometrium in Patients With Repeated IVF Failures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology (Other)
Responsible Party: Principal Investigator, Valeria Muller, PhD, Medical Doctor of Assisted Reproduction Technologies department, D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-001
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infertility, Female; Infertility of Uterine Origin; Asherman Syndrome
Keywords: Repeated IVF failure; Stem cell
MeSH Terms: conditions — Infertility, Female; Gynatresia | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone marrow-derived MSC and HRT (Experimental): endometrial injection of autologous cell product of MSC with hormonal replacement therapy before frozen/thawed ET
  Interventions: Biological: bone marrow-derived MSC and HRT
- hormonal replacement therapy (Active Comparator): standard endometrial preparation for frozen/thawed ET
  Interventions: Other: hormonal replacement therapy

INTERVENTIONS:
Biological: bone marrow-derived MSC and HRT — * Transplantation procedure to endometrial cavity is performed with ultrasound guidance on menstrual cycle day 5-6 through uterine cervix using cater for embryo transfer with 1 ml of suspension containing 5 millions of autologous bone marrow-derived mesenchymal stem cells
  * Three cycles of HRT following MSC transplantation;
  * Pipelle-biopsy of endometrium on day 20 of hormonal replacement therapy of the last (third) cycle;
  * Frozen/thawed embryo transfer 3-6 months after transplantation.
  Arms: bone marrow-derived MSC and HRT
Other: hormonal replacement therapy — standard treatment of hypoplastic endometrium or Asherman's syndrome:
  * Three cycles of HRT preceding frozen/thawed embryo transfer;
  * Frozen/thawed embryo transfer.
  Arms: hormonal replacement therapy

SUMMARY:
Investigators will examine safety and efficiency of the cell product of autologous bone marrow-derived mesenchymal stem cells (MSC) for patients with repeated IVF failures and hypoplastic or/and fibrosis process of endometrium

DETAILED DESCRIPTION:
Sixty patients eligible for the study will be divided to two groups (experimental and control) according to randomization (envelope) procedure in 1:1 ratio.

For patients of the main group bone marrow stem cells will be extracted from the crest of the ilium using standard methodology. After extraction and cultivation final product of autologous bone marrow-derived mesenchymal stem cells will be transplanted to endometrial cavity on menstrual cycle day 5-6. Meanwhile patients will receive three cycles of hormonal replacement therapy (4 mg Progynova (Bayer Pharma, Germany) daily on menstrual cycle day 5-25 in combination with 20 mg Duphaston (Abbott Healthcare Products, B.V., Netherlands) daily from day 15 to day 25. On day 20 of hormonal replacement therapy (HRT) of the last (third) cycle Pipelle-biopsy of endometrium will be performed. Obtained material will be analyzed by immunohistochemistry with the assessment of estrogen and progesterone receptors, VEGFa, GM-CSF, CD133+, CD34 and CD56. Ultrasound characteristics of endometrial quality will be registered on day 9-10 and day 19-21 of every cycle. When morphological and echographic parameters of endometrium are found satisfactory for embryo transfer, the HRT for endometrial preparation for frozen/thawed embryo transfer cycle will be initiated. If acceptable endometrial characteristics are not achieved, patients could be offered to undergo repeated (not more than 3) transplantation of MSC procedures.

Control group will receive three standard cycles of HRT following hysteroscopy before frozen/thawed embryo transfer. If endometrial characteristics are found unsatisfactory, gestational surrogacy might be offered.

ELIGIBILITY:
Inclusion Criteria:

* Repeated IVF attempts with high and good quality embryo transfer in fresh and frozen IVF cycles;
* Age 20-44 years;
* Endometrial thickness less than 6 mm in 2 or more of HRT cycles for endometrial preparation for embryo transfer
* Hysteroscopic evidence of fibrosis processes of uterine cavity with the absence of positive dynamics of HRT in 3 months following operation;
* Signed informed consent.

Exclusion Criteria:

* Contraindication for pregnancy;
* Absence of cryopreserved embryos, stored at clinic's cryobank;
* BMI > 30 kg/m2;
* Impaired carbohydrate metabolism according to glucose tolerance test;
* Thrombosis in anamnesis;
* Oncological diseases in anamnesis;
* Diagnosed inherited thrombophilia;
* Uterine fibroids of more than 4 cm or more than 2 fibroids of 2.5 cm diameter;
* Nodal form of adenomiosis;
* Ovarian cysts more than 4 cm in diameter.

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Assessment of endometrial receptivity | 3-6 month after randomization
  combination of endometrial thickness on ultrasound and immunohistochemistry of endometrium assessed at the biopsy day of the third cycle of HRT

SECONDARY OUTCOMES:
Clinical pregnancy rate | 3-4 weeks after embryo transfer
  presence of intrauterine gestational sac at transvaginal ultrasound at 5-6 weeks of gestation or 5-6 weeks after starting the intervention; measured per frozen/thawed embryo transfer
Treatment-Emergent Adverse Events | 3-6 month after randomization
  Incidence of adverse events: side reactions, abdominal discomfort and patient's tolerance (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Gzgzyan, Prof, PhD, Principal Investigator — D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Locations (1):
- D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No